CLINICAL TRIAL: NCT07001566
Title: The Impact of Cervical Radiculopathy on Functionality and Quality of Life in Patients Undergoing Rotator Cuff Repair
Brief Title: The Impact of Cervical Radiculopathy on Functionality in Patients Undergoing Rotator Cuff Repair
Status: Recruiting | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Assistant Professor, Biruni University
Other Study IDs: Biruni University PTR
Record Dates: First submitted 2025-05-14; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Tears
Keywords: pain; functionality; quality of life
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient's who has cervical radiculopathy: There will be only done assessment.
  Interventions: Other: There was no intervention. Only assessment procedure will be performed.
- Patient's who has not cervical radiculopathy: There will be only done assessment.
  Interventions: Other: There was no intervention. Only assessment procedure will be performed.

INTERVENTIONS:
Other: There was no intervention. Only assessment procedure will be performed. — There was no intervention. Only assessment procedure will be performed.

SUMMARY:
The aim of the study is to evaluate the impact of cervical radiculopathy on functional status and quality of life outcomes in patients who have undergone rotator cuff repair, comparing the group with a history of cervical radiculopathy to the group without cervical radiculopathy.

Study topic: The participants of the study were selected from patients who underwent rotator cuff repair at the Orthopedics and Traumatology clinic of Kartal Dr. Lütfi Kırdar City Hospital between 2018 and 2023. The first group consisted of patients without cervical radiculopathy, while the second group included patients with a previously diagnosed cervical radiculopathy. The study will examine the effect of the presence of cervical radiculopathy on functional outcomes and quality of life in patients who underwent rotator cuff repair.

DETAILED DESCRIPTION:
Shoulder surgery is an important part of modern orthopedic and traumatology practice. Open or closed (arthroscopic) instability and rotator cuff surgeries are the most frequently performed procedures in shoulder surgery.The relationship between cervical spine and rotator cuff pathology has been studied, and the existence of this relationship has been confirmed. Shoulder pain is often associated with rotator cuff tears. Shoulder pain can also result from an external cause, such as cervical radiculopathy. Such a pain source, in conjunction with a rotator cuff tear, can somewhat affect the treatment process of the cuff tear.

Cervical radiculopathy occurs when a nerve root in the spine is compressed or blocked, leading to pain that can radiate beyond the neck, to the arm, chest, shoulders, and upper back. Common symptoms of compression include muscle weakness and impaired deep tendon reflexes. These deficiencies can worsen over time, leading to a decline in quality of life and daily function. While most symptoms can be treated with supportive care, more severe functional loss may require rehabilitation or surgery. Any condition that causes compression or irritation of the spinal nerve root can lead to radicular symptoms. In younger patients, typically in their third and fourth decades, disc trauma and herniation are the most common causes of compression. As age increases, the cause tends to be degenerative. Disc degeneration is the most common cause in the fifth and sixth decades. In the seventh decade, it results from arthritic changes due to foraminal narrowing. Cervical radiculopathies are less frequently seen than lumbar radiculopathies, occurring in approximately 85 per 100,000 people. The C7 nerve root is most frequently affected, with more than half of all cases involving this level. About a quarter of cases involve the C6 nerve root. The C1 to C5 and C8 nerve roots are less affected. Risk factors for developing radicular disease include manual labor such as heavy lifting, driving, or operating vibrating equipment (Magnus, 2024).

Rotator cuff syndrome, also known as rotator cuff tear, is an injury that affects the shoulder, causing pain and inability to use the arm due to the tearing of the muscles and tendons in the rotator cuff. Rotator cuff syndrome can be partial or complete, and is typically caused by injury, trauma, or degeneration. Rotator cuff surgery is rapidly advancing, with most progress driven by improvements in arthroscopic techniques. Generally, functional outcomes are satisfactory. Tendon healing is associated with better results, especially with more strength. Therefore, the best candidates for surgery are those with lesions that have a high likelihood of recovery. Factors associated with recovery include being under 65 years old, having had a recent tear, no history of smoking, having an acromiohumeral distance greater than 6 mm, and a Goutallier fatty degeneration grade of less than 2 in the infraspinatus or subscapularis muscles.

A retrospective cohort study investigated the relationship between cervical spine and rotator cuff pathology and confirmed the existence of this relationship.

In a previous study, it was shown that patients with a history of cervical spine issues who underwent shoulder surgery had lower postoperative functional outcomes, lower satisfaction, and higher rates of postoperative complications requiring surgical revision, compared to patients without cervical spine issues. Another study, focusing on a cohort of patients who underwent shoulder surgery, showed that the short-term postoperative outcomes of patients with cervical spine pathology were significantly lower compared to the functional outcomes of patients without cervical spine pathology.

The sample size was calculated using the G*Power 3.1.9.7 program. The logistic regression test was used, with α error set at 0.20 and 80% power. The odds ratio value from Zhang et al.'s (2015) study, titled The Association Between Cervical Spine Pathology and Rotator Cuff Dysfunction, was used as a reference for patients diagnosed with cervical pathology who developed rotator cuff injury or underwent surgery within a five-year period. Based on this value, the required sample size to achieve 80% power was calculated to be 78 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone rotator cuff repair
* Patients under the age of 65

Exclusion Criteria:

* Patients who have undergone shoulder surgery other than rotator cuff repair
* Patients with a history of cervical spine surgery
* Patients with any neurological disorders
* Patients with a history of pathological fractures
* Patients with oncological diseases
* Patients with a history of infection
* Patients who were deceased at the time of retrospective screening

Ages: 41 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted on 50 patients who underwent rotator cuff surgery between 2018 and 2023, with a mean age of 53.74 ± 6.58 years, 54% of whom were female
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Functionality and quality of life | Between the years 2018 and 2023

SECONDARY OUTCOMES:
pain perception | Between the years 2018 and 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Lütfi Kırdar City Hospital, Istanbul, Istanbul, Turkey (Türkiye)